CLINICAL TRIAL: NCT04330742
Title: The Influence of Intravascular Fluid Administration on Aortic Velocity Time Integral in Obstetric Patients Undergoing Cesarean Section
Brief Title: The Effect of Fluids on Aortic VTI During C-section
Status: Recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Amy Lee, Associate Professor of Obstetric Anesthesiology, Baylor College of Medicine
Other Study IDs: H45744
Record Dates: First submitted 2020-03-28; First posted 2020-04-01 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy Related; Hemorrhage; Fluid Overload; Labor Complication
Keywords: obstetrics; fluid responsiveness; fluid resuscitation
MeSH Terms: conditions — Hemorrhage; Edema; Obstetric Labor Complications | interventions — Ringer's Lactate; Crystalloid Solutions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 0 mL crystalloid: These are the measurements (aortic velocity time integral, inferior vena cava diameter, vital signs) that will be taken at time 0, at which time 0 mL of fluids will have been administered.
  Interventions: Drug: lactated ringers
- 250 mL crystalloid.: These are the measurements (aortic velocity time integral, inferior vena cava diameter, vital signs) that will be taken at time 1, after the spinal has been placed and approximately 250 mL fluids has been administered.
  Interventions: Drug: lactated ringers
- 500 mL crystalloid: These are the measurements (aortic velocity time integral, inferior vena cava diameter, vital signs) that will be taken at time 2, at which time 500 mL of fluids will have been administered.
  Interventions: Drug: lactated ringers
- 1000 mL crystalloid: These are the measurements (aortic velocity time integral, inferior vena cava diameter, vital signs) that will be taken at time 3, at which time 1000 mL of fluids will have been administered.
  Interventions: Drug: lactated ringers

INTERVENTIONS:
Drug: lactated ringers — the intervention is one liter fluid bag of lactated ringers which is routinely used as a fluid coload for spinal anesthesia. All patients will receive the same amount of fluids however this will be paused at various time points in order to perform the echocardiogram.
  Other Names: crystalloid

SUMMARY:
Pregnancy is associated with a myriad of physiologic changes, including expansion of blood volume, decrease in oncotic pressure, and increased cardiac output. The obstetric population is associated with intrapartum hemorrhage. Accordingly, it is important to have an accurate method to assess fluid status in intrapartum patients. The use of standard volume assessment tools including arterial lines and central venous catheters is limited given the brevity of obstetric procedures and the morbidity of these techniques on the awake patients, and the costs. Non-invasive methods to assess volume status (carotid dopplers, direct measurement of blood loss, bio-impedance devices) are imperfect. Echocardiography is an attractive tool to measure fluid status in experienced operators such as anesthesiologists. IVC diameter and variation of aortic velocity time integral are two measures that can be obtained via echocardiography and been studied in spontaneously breathing patients. The purpose of this study is to determine whether these measurements can be used in the assessment of volume status in the laboring patient.

DETAILED DESCRIPTION:
Pregnancy is associated with a myriad of physiologic changes, including expansion of blood volume, decrease in oncotic pressure, and increased cardiac output. Comorbidities including maternal hypertension, renal or cardiac disease may further complicate the assessment of volume status and are associated with increased risks related to fluid administration (c). In addition, the majority of obstetric patients receive neuraxial analgesia or anesthesia to facilitate both vaginal and operative delivery. These techniques are associated with hemodynamic changes including maternal hypotension secondary to a decrease in SVR and CO. These changes may in turn be associated with a reduction in placental blood flow affecting fetal outcome, and may also cause maternal nausea, vomiting and dizziness. Further, the obstetric population is high risk for intrapartum hemorrhage. As such, it is critical to have an accurate method to assess fluid status in intrapartum patients.

The use of invasive volume assessment tools including arterial lines and central venous catheters is limited given the brevity of obstetric procedures, the morbidity of these invasive techniques for the awake patient, and the associated time and costs (b). Non-invasive methods that assess volume status in the obstetric population include techniques such as direct measurement of blood loss (g), carotid dopplers (c), bio-impedence devices (f); However these methods have been shown to be imperfect and are not widely used.

Echocardiography is a non-invasive, widely-available tool that can provide rapid information for experienced operators such as anesthesiologists. Respiratory variations in inferior vena cava diameter (IVCd) and variation in aortic velocity time integral (∆VTI) following passive leg raise have been extensively studied in spontaneously breathing patients. IVCd has been shown to predict fluid responsiveness, however requires a high threshold (>40-50% collapsibility) to detect a difference. IVCd may also change with diaphragmatic motion, thus results may be confounded if the patient becomes tachypneic (d) or is spontaneously breathing (g). In contrast, aortic velocity time integral (∆VTI) may be a more sensitive indicator of volume status. Lamia et al showed a 12% change in VTI as 77% sensitive and 100% specific for a 15% change in cardiac output following 500 mL volume expansion in ICU patients with shock (both spontaneously breathing and mechanically ventilated, e). While there are some studies of IVC collapsibility in the obstetric population, there are limited data on VTI as a measure of volume status in laboring patients.

The purpose of this study is to determine whether the aortic velocity time integral (VTI) is influenced by intravascular fluid administration during cesarean section. Secondary aims include determining whether inferior vena cava diameter (IVCd), blood pressure, and heart rate are influenced by intravascular fluid administration during cesarean section. Additionally, total amount of vasopressor agents administered during the procedure will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* healthy nulliparous or multiparous pregnant women with a term (>37 weeks gestation)
* age 18-35
* singleton pregnancy
* scheduled for Cesarean delivery with planned neuraxial spinal or combined spinal epidural anesthesia
* American Society for Anesthesiologists physical status 2

Exclusion Criteria:

* Patients without ability to provide informed consent
* American Society for Anesthesiologists physical status 3 or 4
* Emergency cesarean section
* BMI>40
* Known cardiac and pulmonary comorbidities including chronic hypertension, preeclampsia, gestational hypertension, diabetes, asthma, renal disease
* Age > 35

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients ages 18-35 undergoing elective cesarean section with planned spinal anesthetic at Ben Taub General Hospital (BTGH) will be screened. Consenting patients will undergo spinal anesthetic prior to planned procedure. All subjects will receive the same 1L fluid bolus intraoperatively.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-03-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
aortic velocity time integral | at baseline measure, right after spinal placement (250mL LR), at 500mL LR infusion, and at 1 L LR infusion (approximately 20mins)
  the percent change in aortic velocity time integral as measured by transthoracic echo

SECONDARY OUTCOMES:
inferior vena cava collapsibility | at baseline measure, right after spinal placement (250mL LR), at 500mL LR infusion, and at 1 L LR infusion (approximately 20mins)
  the percent change in diameter of inferior vena cava as measured by transthoracic echo
change in systolic blood pressure | every 2.5 mins for 20 mins (when 1L LR is administered) once the pt has a spinal placement
  percent change in systolic blood pressure
change in heart rate | every 2.5 mins for 20 mins (when 1L LR is administered) once the pt has a spinal placement
  percent change in heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Amy Lee, MD, Principal Investigator — Baylor College of Medicine; Yi Deng, MD, Study Director — Baylor College of Medicine; Claudia Wei, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Ben Taub General Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ngan Kee WD, Khaw KS, Ng FF. Prevention of hypotension during spinal anesthesia for cesarean delivery: an effective technique using combination phenylephrine infusion and crystalloid cohydration. Anesthesiology. 2005 Oct;103(4):744-50. doi: 10.1097/00000542-200510000-00012. PMID 16192766
- [Background] Zieleskiewicz L, Noel A, Duclos G, Haddam M, Delmas A, Bechis C, Loundou A, Blanc J, Mignon A, Bouvet L, Einav S, Bourgoin A, Leone M. Can point-of-care ultrasound predict spinal hypotension during caesarean section? A prospective observational study. Anaesthesia. 2018 Jan;73(1):15-22. doi: 10.1111/anae.14063. Epub 2017 Oct 7. PMID 28986931
- [Background] Zieleskiewicz L, Bouvet L, Einav S, Duclos G, Leone M. Diagnostic point-of-care ultrasound: applications in obstetric anaesthetic management. Anaesthesia. 2018 Oct;73(10):1265-1279. doi: 10.1111/anae.14354. Epub 2018 Jul 26. PMID 30047997
- [Background] Lamia B, Ochagavia A, Monnet X, Chemla D, Richard C, Teboul JL. Echocardiographic prediction of volume responsiveness in critically ill patients with spontaneously breathing activity. Intensive Care Med. 2007 Jul;33(7):1125-1132. doi: 10.1007/s00134-007-0646-7. Epub 2007 May 17. PMID 17508199
- [Background] McIntyre JP, Ellyett KM, Mitchell EA, Quill GM, Thompson JM, Stewart AW, Doughty RN, Stone PR; Maternal Sleep in Pregnancy Study Group. Validation of thoracic impedance cardiography by echocardiography in healthy late pregnancy. BMC Pregnancy Childbirth. 2015 Mar 28;15:70. doi: 10.1186/s12884-015-0504-5. PMID 25886289
- [Background] Hancock A, Weeks AD, Lavender DT. Is accurate and reliable blood loss estimation the 'crucial step' in early detection of postpartum haemorrhage: an integrative review of the literature. BMC Pregnancy Childbirth. 2015 Sep 28;15:230. doi: 10.1186/s12884-015-0653-6. PMID 26415952
- [Background] Airapetian N, Maizel J, Alyamani O, Mahjoub Y, Lorne E, Levrard M, Ammenouche N, Seydi A, Tinturier F, Lobjoie E, Dupont H, Slama M. Does inferior vena cava respiratory variability predict fluid responsiveness in spontaneously breathing patients? Crit Care. 2015 Nov 13;19:400. doi: 10.1186/s13054-015-1100-9. PMID 26563768
- [Background] Brun C, Zieleskiewicz L, Textoris J, Muller L, Bellefleur JP, Antonini F, Tourret M, Ortega D, Vellin A, Lefrant JY, Boubli L, Bretelle F, Martin C, Leone M. Prediction of fluid responsiveness in severe preeclamptic patients with oliguria. Intensive Care Med. 2013 Apr;39(4):593-600. doi: 10.1007/s00134-012-2770-2. Epub 2012 Dec 6. PMID 23223774
- [Background] Muller L, Bobbia X, Toumi M, Louart G, Molinari N, Ragonnet B, Quintard H, Leone M, Zoric L, Lefrant JY; AzuRea group. Respiratory variations of inferior vena cava diameter to predict fluid responsiveness in spontaneously breathing patients with acute circulatory failure: need for a cautious use. Crit Care. 2012 Oct 8;16(5):R188. doi: 10.1186/cc11672. PMID 23043910
- [Background] Maizel J, Airapetian N, Lorne E, Tribouilloy C, Massy Z, Slama M. Diagnosis of central hypovolemia by using passive leg raising. Intensive Care Med. 2007 Jul;33(7):1133-1138. doi: 10.1007/s00134-007-0642-y. Epub 2007 May 17. PMID 17508202
- [Background] Gardin JM, Davidson DM, Rohan MK, Butman S, Knoll M, Garcia R, Dubria S, Gardin SK, Henry WL. Relationship between age, body size, gender, and blood pressure and Doppler flow measurements in the aorta and pulmonary artery. Am Heart J. 1987 Jan;113(1):101-9. doi: 10.1016/0002-8703(87)90016-0. PMID 2948377
- [Background] Tawfik MM, Tarbay AI, Elaidy AM, Awad KA, Ezz HM, Tolba MA. Combined Colloid Preload and Crystalloid Coload Versus Crystalloid Coload During Spinal Anesthesia for Cesarean Delivery: A Randomized Controlled Trial. Anesth Analg. 2019 Feb;128(2):304-312. doi: 10.1213/ANE.0000000000003306. PMID 29461392
- [Background] Practice Guidelines for Obstetric Anesthesia: An Updated Report by the American Society of Anesthesiologists Task Force on Obstetric Anesthesia and the Society for Obstetric Anesthesia and Perinatology. Anesthesiology. 2016 Feb;124(2):270-300. doi: 10.1097/ALN.0000000000000935. No abstract available. PMID 26580836